CLINICAL TRIAL: NCT02950155
Title: A Randomized, Double-blind, Placebo-controlled Multicenter Study Evaluating the Safety and Efficacy of Rituximab (Mabthera®) in Patients With New Onset Generalized Myasthenia Gravis (MG)
Brief Title: A Study Evaluating the Safety and Efficacy of Rituximab in Patients With Myasthenia Gravis
Acronym: Rinomax
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fredrik Piehl (Other)
Responsible Party: Sponsor-Investigator, Fredrik Piehl, Professor, MD, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EudraCT 2015-005749-30
Record Dates: First submitted 2016-10-28; First posted 2016-10-31 (Estimated); Results first posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-08

CONDITIONS: Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Rituximab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Experimental): A single infusion at a dose of 500 mg of Mabthera/Rituximab.
  Interventions: Drug: Rituximab
- Sodium Chloride solution (Sham Comparator): A single infusion with sodium chloride solution.
  Interventions: Drug: Sodium Chloride solution

INTERVENTIONS:
Drug: Rituximab — A single infusion at a dose of 500 mg Mabthera/Rituximab.
  Other Names: Mabthera
  Arms: Rituximab
Drug: Sodium Chloride solution — A single infusion of Placebo/Sham.
  Other Names: Sodium Chloride
  Arms: Sodium Chloride solution

SUMMARY:
A randomized, double-blind, placebo-controlled multicenter study evaluating the safety and efficacy of Rituximab (Mabthera®) in patients with new onset generalized myasthenia gravis (MG).

DETAILED DESCRIPTION:
Myasthenia gravis (MG) is an autoimmune disease of the neuromuscular junction caused by auto-antibodies. MG is characterized by weakness in skeletal muscles and occurs in all ages, but mostly among young adult women and in people of both sexes over the age of 60 years. The disease has a wide variation in severity, where in milder cases only symptom-relieving choline esterase blockers may be sufficient. In many cases, however, immunomodulatory drugs are required. Traditionally MG has been treated with high doses of corticosteroids over longer time periods, which causes significant risks of side effects. Therefore, since several decades, oral immunosuppressive drugs have been used in order to reduce the need for steroids. This group includes azathioprine, cyclosporine and mycophenolate. However, none of these drugs has been approved for use in MG and the effect is usually delayed. There is thus a great need to develop newer treatment algorithms for MG, for example including more effective biological drugs. Several small observational studies have shown that rituximab, an anti-CD20 monoclonal antibody that eliminate B cells, can have good effects in treatment refractory MG. The aim of the present study is to study the effect of rituximab compared to placebo in the treatment of new onset MG of moderate to severe symptomatology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with oculobulbar, bulbar or generalized MG ≥ 18 years of age and with onset of generalized symptoms or neurophysiological detection of generalized disease not more than 12 months ago.
2. The diagnosis of MG should be determined with the following:

   Clinical neurological status with motor symptoms consistent with MG and at least two of the following:

   a positive serologic test for anti-acetylcholine receptor antibody (AChR) and/or b. typical MG findings on neurophysiological testing of neuromuscular transmission with single fiber electromyography (SFEMG) and / or repetitive nerve stimulation (RNS), and / or c. Positive anti-choline esterase-test, e.g. edrophoniumchloride or improvement of MG symptoms with oral cholinesterase inhibitors as judged by the treating physician.
3. MGFA Class II to IV at screening.
4. Quantitative MG score ≥ 6 at screening
5. Women of childbearing potential must have a negative pregnancy test.
6. Patients must have provided written informed consent.
7. Patients must be able and willing to comply with all study procedures.

Exclusion Criteria:

1. Weakness only affecting ocular or periocular muscles (MGFA Class I).
2. MG crisis at screening (MGFA Class V)
3. Thymectomy already carried out. In order to avoid difficulties to evaluate the effect of the study drug, thymectomy, where it is indicated, should be scheduled to the follow-up period, ie after the first 24 weeks.
4. Strong suspicion of thymoma, where thymectomy as judged by the treating physician should be done within 24 weeks.
5. Active malignancy, if not adequately treated
6. Pregnancy or breast-feeding.
7. Ongoing acute or chronic viral or systemic bacterial infections including HIV, latent hepatitis B, which is clinically significant, according to the study doctor's opinion and not treated with appropriate antibiotic / antiviral drugs.
8. Severe heart failure (New York Heart Association Class IV) or severe, uncontrolled cardiac disease
9. Previous use of immunosuppressive drugs, including rituximab, except prednisolone at a dose of up to 40mg daily for less than 3 months. This does not apply to treatment with immunosuppressive drugs / corticosteroids (except rituximab) for other indications than MG, provided at least 12 months have passed since treatment was terminated.
10. Suspected hypersensitivity to the study drug
11. Participation in another trial of study drug within 30 days prior to screening.
12. Any medical condition which, according to the study physician's opinion, may interfere with the patient's participation in the study, poses additional risks for the patient, or that complicate the assessment of patients.
13. Vaccination within 4 weeks before inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-10-16 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Piehl, Professor, Principal Investigator — Dept Clinical Neuroscience Karolinska Institutet, Neuroimmunology Unit
Locations (1):
- Karolinska University Hospital, Stockholm, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piehl F, Eriksson-Dufva A, Budzianowska A, Feresiadou A, Hansson W, Hietala MA, Hakansson I, Johansson R, Jons D, Kmezic I, Lindberg C, Lindh J, Lundin F, Nygren I, Punga AR, Press R, Samuelsson K, Sundstrom P, Wickberg O, Brauner S, Frisell T. Efficacy and Safety of Rituximab for New-Onset Generalized Myasthenia Gravis: The RINOMAX Randomized Clinical Trial. JAMA Neurol. 2022 Nov 1;79(11):1105-1112. doi: 10.1001/jamaneurol.2022.2887. PMID 36121672

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 16th, 2016, and March 2nd, 2020, 87 potentially eligible patients were screened at 7 Swedish neurology clinics (5 university hospitals, 2 regional hospitals). 47 fulfilled inclusion and exclusion criteria and provided informed consent to participation.
Pre-assignment Details: All included participants received study drug
Groups:
- Rituximab: A single intravenous infusion at a dose of 500 mg of Mabthera/Rituximab in Sodium Chloride solution.
- Placebo: A single intravenous infusion with sodium chloride solution in infusion bag matched to active treatment.
Period: Overall Study
Arm/Group | Rituximab | Placebo
Started | 25 | 22
Completed | 25 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Rituximab: A single infusion at a dose of 500 mg of Mabthera/Rituximab in Sodium Chloride solution.
- Sodium Chloride Solution: A single infusion with sodium chloride solution in infusion bag matched to active treatment.
- Total: Total of all reporting groups
Arm/Group | Rituximab | Sodium Chloride Solution | Total
Number analyzed (Participants) | 25 | 22 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (13.4) | 58.0 (18.6) | 63.0 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 18 | 15 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 25 | 22 | 47
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.5 (3.7) | 27.6 (5.7) | 27.5 (4.7)
Concentration of acetylcholine receptor antibodies [Mean (Standard Deviation); unit: nmol/L] | 22.7 (19.3) | 70.7 (117) | 46.7 (86.5)
Time since onset of generalized symptoms of myasthenia gravis [Mean (Standard Deviation); unit: days] | 132.4 (91.5) | 143.0 (93.3) | 137.4 (91.5)
Ocular symptoms prior to generalized symptoms of myasthenia gravis [Number; unit: participants] | 4 | 2 | 6
Quantitative Myasthenia Gravis score [Mean (Standard Deviation); unit: units on a scale] — The Quantitative Myasthenia Gravis (QMG) score is a physician rated disease activity score which ranges from 0 (minimum) to 39 (maximum) units on the scale. Lower score indicates better outcome.
  units on a scale | 9.4 (4.5) | 9.3 (4.5) | 9.4 (4.4)
Myasthenia Gravis Quality of Life questionnaire score [Mean (Standard Deviation); unit: units on a scale] — The Myasthenia Gravis Quality of Life (MG-QoL) questionnaire is a patient rated quality of life score which ranges from 0 (minimum) to 60 (maximum) units on the scale. Lower score indicates better outcome.
  units on a scale | 20.1 (11.0) | 22.2 (12.8) | 21.1 (11.8)
Myasthenia Gravis Activities of Daily Living score [Mean (Standard Deviation); unit: units on a scale] — The Myasthenia Gravis Activities of Daily Living (MG-ADL) scale is a patient rated disease activity score which ranges from 0 (minimum) to 24 (maximum) units on the scale. Lower score indicates better outcome.
  units on a scale | 5.1 (3.2) | 4.5 (2.7) | 4.9 (2.9)
Prednisolone [Count of Participants; unit: Participants] — Number of patients treated with oral Prednisolone at baseline.
  Participants | 16 | 12 | 28
Dose of Prednisolone (mg/day) [Mean (Standard Deviation); unit: mg/day] — Average daily dose Prednisolone for the above indicated patients treated with oral Prednisolone at baseline. Population: Average daily dose of Prednisolone for patients treated at baseline.
  mg/day
    number analyzed (Participants) | 16 | 12 | 28
    (all) | 22.5 (10.8) | 20.8 (9.0) | 21.8 (9.9)
Intravenous immunoglobulins prior to baseline [Count of Participants; unit: Participants] — Number of patients treated with intravenous immunoglobulins (IVIG) within three months prior to baseline.
  Participants | 8 | 8 | 16
Plasmapheresis prior to baseline [Count of Participants; unit: Participants] — Number of patients treated with Plasmapheresis (PLEX) within three months prior to baseline.
  Participants | 1 | 0 | 1
Early-onset myasthenia gravis [Count of Participants; unit: Participants] — Subgroup defined as anti-AChR+ and age <50 years at onset
  Participants | 2 | 7 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Quantitative MG Score (QMG) Score ≤ 4 and a Daily Prednisolon Dose of ≤ 10mg at 16 Weeks After Administration of Study Drug/Placebo.
Description: The Quantitative Myasthenia Gravis (QMG) score is a physician rated disease activity score that ranges from 0 to 39, where lower indicates better outcome. QMG was measured at 16 weeks under standardized conditions with at least 12 hours since last intake of choline esterase inhibitors. Patients meeting the primary outcome had a QMG score of 4 or less whilst also requiring a daily oral Prednisolone dose of 10 mg or less.
Time Frame: 16 weeks
Population: Missing data, rituximab=1, placebo=1
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Sodium Chloride Solution
Number analyzed (Participants) | 24 | 21
Participants | 17 | 6
Statistical Analysis 1: Comparison: Rituximab vs Sodium Chloride Solution; The primary end-point was analyzed as an intention-to-treat analysis, with Fisher's exact test of the difference in proportion, with α=0·05 to indicate statistically significant difference; Test type: Superiority; p = 0.007, Fisher Exact; probability ratio = 2.48, 95% CI 2-sided [1.20 to 5.11]

2. Secondary Outcome: Change in QMG Score From Week 0 to Week 24 After Administration of Study Drug/Placebo.
Description: The Quantitative Myasthenia Gravis (QMG) score is a physician rated disease activity score that ranges from 0 to 39, where lower indicates better outcome. QMG was measured under standardized conditions with at least 12 hours since last intake of choline esterase inhibitors. Change in QMG scores between the two time points was compared between groups.
Time Frame: 24 weeks
Population: censured patients, rituximab=2, placebo=9
Measure: Mean (Standard Deviation); unit: change in score points
Arm/Group | Rituximab | Sodium Chloride Solution
Number analyzed (Participants) | 23 | 13
change in score points | -6.9 (5.6) | -5.8 (4.6)
Statistical Analysis 1: Comparison: Rituximab vs Sodium Chloride Solution; Subjects receiving rescue treatment before evaluation being censored (per-protocol analysis); Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-4.4 to 2.1]

3. Secondary Outcome: Change in Myasthenia Gravis Activities of Daily Living (MG-ADL) Score From Week 0 to Week 16 After Administration of Study Drug/Placebo
Description: The Myasthenia Gravis Activities of Daily Living (MG-ADL) score is a patient rated disease activity score that ranges from 0 to 24, where lower indicates better outcome. MG-ADL was assessed at 16 weeks under standardized conditions with at least 12 hours since last intake of choline esterase inhibitors. Change in MG-ADL scores between the two time points was compared between groups.
Time Frame: 16 weeks
Population: censured patients, rituximab=3, placebo=7
Measure: Mean (Standard Deviation); unit: change in score points
Arm/Group | Rituximab | Sodium Chloride Solution
Number analyzed (Participants) | 22 | 15
change in score points | -1.7 (2.5) | -0.5 (3.6)
Statistical Analysis 1: Comparison: Rituximab vs Sodium Chloride Solution; Subjects receiving rescue treatment before evaluation being censored (per-protocol analysis); Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-3.3 to 0.8]

4. Secondary Outcome: Change in Myasthenia Gravis Quality of Life (QoL) Score From Week 0 to Week 16 After Administration of Study Drug/Placebo.
Description: The Myasthenia Quality of Life (QoL) score is a patient rated quality of life score that ranges from 0 to 60, where lower indicates better outcome. Change in MG-QoL scores between the two time points was compared between groups.
  .
Time Frame: 16 weeks
Population: censured patients, rituximab=3, placebo=7
Measure: Mean (Standard Deviation); unit: change in score points
Arm/Group | Rituximab | Sodium Chloride Solution
Number analyzed (Participants) | 22 | 15
change in score points | -9.2 (9.2) | -7.0 (9.3)
Statistical Analysis 1: Comparison: Rituximab vs Sodium Chloride Solution; Subjects receiving rescue treatment before evaluation being censored (per-protocol analysis); Test type: Superiority; p = 0.47, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-8.2 to 3.8]

5. Other Pre Specified Outcome: Percentage of Patients With Quantitative MG Ascore (QMG) Score ≤ 4 and a Daily Prednisolon Dose of ≤ 10mg at 24 Weeks After Administration of Study Drug/Placebo.
Description: The Quantitative Myasthenia Gravis (QMG) score is a physician rated disease activity score that ranges from 0 to 39, where lower indicates better outcome. QMG was measured at 24 weeks under standardized conditions with at least 12 hours since last intake of choline esterase inhibitors. Patients meeting the primary outcome had a QMG score of 4 or less whilst also requiring a daily oral Prednisolone dose of 10 mg or less.
Time Frame: 24 weeks
Population: missing data, rituximab=0, placebo=1
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Sodium Chloride Solution
Number analyzed (Participants) | 25 | 21
Participants | 18 | 8
Statistical Analysis 1: Comparison: Rituximab vs Sodium Chloride Solution; Test type: Superiority; p = 0.036, Fisher Exact; probability ratio = 1.89, 95% CI 2-sided [1.04 to 3.44]

6. Other Pre Specified Outcome: QMG Scores at 16, 36 and 48 Weeks After Administration of Study Drug/Placebo.
Description: QMG is measured under standardized conditions with at least 12 hours since last intake of choline esterase inhibitors
Time Frame: 16, 36 and 48 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: MG-activities of Daily Living (ADL) Score at 24, 36 and 48 Weeks After Administration of Study Drug/Placebo
Description: MG-ADL is a patient-reported outcome measured under standardized conditions with at least 12 hours since last intake of choline esterase inhibitors
Time Frame: 24, 36 and 48 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: EQ5D Score at 16, 24, 36 and 48 Weeks After Administration of Study Drug/Placebo
Description: The EQ5D scale is a generic QoL score measured under standardized conditions with at least 12 hours since last intake of choline e
Time Frame: 16, 24, 36 and 48 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: MG-QoL Score at 24, 36 and 48 Weeks After Administration of Study Drug/Placebo
Description: MG-QoL is a patient-reported outcome measured under standardized conditions with at least 12 hours since last intake of choline esterase inhibitors
Time Frame: 24, 36 and 48 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Number of Hospital Admissions for MG Worsening During Week 0 to 24 After Administration of Study Drug/Placebo
Description: The total number of hospital admissions for MG worsening during week 0 to 24 of the study.
Time Frame: 24 weeks
Measure: Number; unit: hospital adminssions
Groups:
- Placebo: A single infusion with sodium chloride solution in infusion bag matched to active treatment.
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 25 | 22
hospital adminssions | 0 | 3

11. Other Pre Specified Outcome: Rescue Treatments During Week 8 to 24 After Administration of Study Drug/Placebo
Description: The number of events when rescue treatment was given during week 8-24 of the study. Rescue treatments were defined as i.v immunoglobulins, plasma exchange, high dose corticosteroids and biologics (rituximab, tocilizumab).
Time Frame: 8 - 24 weeks
Measure: Number; unit: events
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 25 | 22
events | 1 | 8

ADVERSE EVENTS:
Time Frame: 48 weeks, i.e. time from baseline to last follow up.
Description: The definitions described in clinicaltrials.gov are used with no exception. Information on potential adverse events was collected at each study visit (n=5) and telephone follow-ups (n=4).
Arm/Group | Rituximab | Sodium Chloride Solution
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/22
Serious Adverse Events (participants affected / at risk) | 5/25 | 4/22
Other Adverse Events (participants affected / at risk) | 21/25 | 17/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=25) | Sodium Chloride Solution (N=22)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Septicaemia (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Nervous system disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 2 (2) | 0 (0)
Asystole (Cardiac disorders) | 0 (0) | 1 (2)
Vertebral compression fracture (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Syncope (Cardiac disorders) | 1 (1) | 0 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=25) | Sodium Chloride Solution (N=22)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Allergic reaction (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Arrythmia (Cardiac disorders) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 6 (7) | 8 (10)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0)
Fever of unknown cause (Infections and infestations) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Rectal bleeding (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 4 (4)
Urine leaks (Renal and urinary disorders) | 2 (2) | 1 (1)
Kidney stone (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary tract infection (Renal and urinary disorders) | 2 (3) | 0 (0)
Bite from animal (dog) (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Imbalances in some baseline characteristics, with a lower age, higher AChR antibody titres, a lower proportion treated with prednisolone, and a greater proportion with MGFA class III disease among those randomized to placebo compared with rituximab. On the other hand, late onset MG has been associated with worse disease, and one subject in the active arm suffered a condition (ALS) that effectively excluded the possibility to evaluate a treatment effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT02950155/Prot_SAP_000.pdf